CLINICAL TRIAL: NCT02669290
Title: Use of 3-D Blood Pool Scintigraphy to Guide Left Ventricular Pacing Lead Placement in Patients Requiring Cardiac Resynchronization Therapy (MUGA-CRT)
Brief Title: Use of 3-D Blood Pool Scintigraphy to Guide Left Ventricular Pacing Lead Placement in Patients Requiring Cardiac Resynchronization Therapy
Acronym: MUGA CRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-04791
Record Dates: First submitted 2016-01-13; First posted 2016-02-01 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Left Ventricular Dysfunction; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided (Experimental): Guided LV lead placement for CRT.
  Interventions: Other: Guided
- Non-Guided (Active Comparator): Non-guided LV lead placement for CRT.
  Interventions: Other: Non-guided

INTERVENTIONS:
Other: Guided — LV lead placement will be guided by left ventricular systolic function information from MUGA
  Arms: Guided
Other: Non-guided — LV lead placement will be conventional posterolateral placement
  Arms: Non-Guided

SUMMARY:
The purpose of this study is to determine whether multiple gated acquisition (MUGA) guided lead placement improves clinical outcomes for patients needing cardiac resynchronization therapy (CRT) compared to traditional posterolateral left ventricular lead placement.

DETAILED DESCRIPTION:
Heart failure (HF) has a prevalence of five million individuals in the United States. Approximately 25-30% of patients with HF due to left ventricular (LV) systolic dysfunction have prolonged QRS. Prolonged QRS duration (>120ms) on ECG in HF patients is associated with increased morbidity and mortality.

Delayed electrical activation of the LV translates to temporal delay in ventricular contraction. This is referred to as mechanical dyssynchrony. Patients with advanced HF, low ejection fraction (EF) of less than 35% and QRS of more than 120ms are indicated for cardiac resynchronization therapy (CRT). While most patients undergoing CRT implantation show dramatic improvement in HF symptoms, 30-40% of the HF patients undergoing CRT placement do not show a clinical response. The site of placement of the LV lead has been shown to be an important determinant of the effects of CRT.

Measurement of left ventricular ejection fraction (LVEF) is performed using non-invasive measures such as the MUGA. By using the available information on left ventricular systolic function the investigators plan on investigating the effects of MUGA-guided versus traditional LV lead placement for CRT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Must have an approved indication for CRT implantation
* Must have ischemic or nonischemic dilated cardiomyopathy
* Must have symptomatic HF with a New York Association (NYHA) Classification of III or IV
* Must be on optimal pharmacological therapy (this should include at the minimum, ACE inhibitor and beta-blocker therapy as tolerated.
* Must have left ventricular ejection fraction (LVEF) of ≤35%
* Must have ventricular conduction delay manifested as a QRS duration of >120msec
* Must be able to provide informed consent for study participation and be willing to comply with follow-up tests and scheduled visits

Exclusion Criteria:

* HF diagnosis for less than 3 months
* Physical limitations to ambulation
* Life expectancy of less than six months
* Pregnant or planning for pregnancy in the next 6 months (must have a negative pregnancy test 7 days prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Six minute walk test (6MWT) | Baseline to six months.
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.

SECONDARY OUTCOMES:
Change in New York Heart Association (NYHA) class. | Baseline to six months.
  Clinicians classify patients' heart failure according to the severity of their symptoms.
Quality-of-Life Questionnaire | Baseline to six months.
  Minnesota Living with Heart Failure Questionnaire: To measure the effects of symptoms, functional limitations, psychological distress on an individual's quality of life, the MLHF questionnaire asks each person to indicate using a 6-point, zero to five, Likert scale how much each of 21 facets prevented them from living as they desired.
Echocardiogram (echo) Parameters | Baseline to six months.
  Echo is a type of ultrasound test that takes pictures of the heart. These pictures will be used to assess whether there are any improvements in left ventricular function.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided